CLINICAL TRIAL: NCT03264170
Title: Implementation of a Model for Predicting Early Pregnancy Outcome in Women With Pregnancy of Uncertain Viability: a Psychological Impact Study
Brief Title: Psychological Impact of Predicting Early Pregnancy Outcomes in Women With Pregnancy of Uncertain Viability
Acronym: IMPROVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: C&W17/082017
Record Dates: First submitted 2017-08-21; First posted 2017-08-29 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2017-08

CONDITIONS: Uncertain Viability of Pregnancy; Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: All participating women will be randomised to one of two groups at the time of recruitment. The intervention group will receive the prediction score. The control group will not receive the prediction score.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prediction of pregnancy outcome (Active Comparator): Women will receive an individualised prediction score of the pregnancy being viable at the follow-up ultrasound generated from the prediction tool.
  Interventions: Diagnostic Test: Prediction of pregnancy outcome
- Control (No Intervention): Women will not receive the prediction score

INTERVENTIONS:
Diagnostic Test: Prediction of pregnancy outcome — The intervention group will receive the individualised prediction of their pregnancy (as a percentage). The prediction is calculated by a validated, accurate mathematical model using specific background information and ultrasound data for each participant.
  Arms: Prediction of pregnancy outcome

SUMMARY:
This study will evaluate if providing women diagnosed with an intrauterine pregnancy of uncertain viability with a percentage likelihood of ongoing viability of their pregnancy at the time of the follow-up ultrasound, will result in improved psychological well-being (reduced anxiety and depression). Recruited women will be randomised to either receive the prediction score (intervention arm) or not (control arm).

DETAILED DESCRIPTION:
Intrauterine pregnancy of uncertain viability (IPUVI) affects 10-28% of women seen in the Early Pregnancy Assessment Unit (EPAU). Such women have a pregnancy correctly sited within the uterus but the viability of the pregnancy cannot be determined at the initial scan. This finding may represent a normally developing (but early) pregnancy. However, approximately 50% of these pregnancies will eventually miscarry. The current recommendation from The National Institute for Health and Care Excellence (NICE) is to offer a confirmatory scan after 14 days.

This 14-day interval is particularly distressing for women and diagnostic uncertainty in early pregnancy is associated with heightened levels of anxiety and depression. NICE Evidence Update 71 (2014) suggests that provision of more information about the likely outcome of the pregnancy (prior to the repeat ultrasound) may benefit psychological health.

The investigators have previously developed, validated and published a mathematical tool to predict pregnancy viability after diagnosis of IPUVI (549 participants). The tool (which takes account of maternal age, vaginal bleeding score and ultrasound measurements) is established as an accurate research tool having been externally validated in a different test population. Having established its performance, the investigators would like to provide women with this individualised prediction of their pregnancy outcome. If psychologically beneficial (and not harmful) this tool may help up to a third of the EPAU population.

This will be a single centre, prospective non-blind randomised control study. All eligible women with IPUVI ultrasound classification at Chelsea and Westminster Hospital will be identified and invited to be recruited to the study.

Following recruitment, a woman will be randomised by random computer generator to either Group I (intervention group - receive the prediction score) or Group II (control group - do not receive the prediction score).

Potential participants will be identified on a daily basis by those that regularly perform ultrasound scans within the department; sonographers, nurse specialists, research fellows and consultants. Once identified, they shall be approached by the local researcher for a face-to-face consultation who will confirm their eligibility criteria and explain the study. In addition, the detailed patient information sheet (PIS) will be provided before taking informed written consent. Clinicians who perform ultrasound scans out of hours, will be notified of the study and asked to inform eligible women about the study and obtain consent for the local researcher to contact them the next working day.

Written, informed consent will be taken prior to recruitment from all participants. It will clearly state that the participant is free to withdraw from the study at any time for any reason without prejudice to future care, and with no obligation to give the reason for withdrawal.

It is estimated that a total of 250 women will be recruited (125 participants in each group). Data will be collected from all women at three points during the course of the study. A single, validated scale will be used for data collection regarding psychological well-being. The questionnaire to be used is the Hospital Anxiety and Depression Scale (HADS) by Zigmond and Snaith (1983).

Each questionnaire will take approximately 5-10 minutes to complete. The questionnaires will be sent to participants via email (or post if participants do not have access to email). If a participant does not initially respond the researcher may send one reminder email and contact them by telephone on one occasion with prior consent from the participant. If the participant does not respond following these reminders they will be withdrawn from the study. The local researcher will monitor the progress of each participant's pregnancy prior to sending out the questionnaires. Women who are known to have undergone termination of pregnancy prior to completion of all three questionnaires will be withdrawn from the study and not contacted with further questionnaires.

Participants in Group I will also be invited to complete a patient experience questionnaire at the end of the study period to assess their perceived acceptability and usefulness of the tool. This has been developed specifically for this study using modified versions of the Technology Acceptance Model (Davis et al 1989).

The potential benefits of the study are outlined. This study will confirm whether this prediction tool is of clinical and psychological benefit to the patient.

Women may find the questionnaires they are asked to complete prompt them to seek help earlier for conditions which may otherwise have gone untreated such as anxiety and depression. In addition, they may find it therapeutic to be able to express their opinions, emotions and feelings during the period of uncertainty.

If the study shows that the prediction tool is acceptable to patients (as well as being accurate in terms of the actual pregnancy outcome) this will allow units to more appropriately triage follow-up plans were resources are limited.

Following the study, it is anticipated that the use of the tool could be extended to other clinical sites to aid the management and expectations of women diagnosed with IPUVI. The NICE Evidence Update specifically refers to this prediction tool and it is anticipated that this will be a nationally recommended tool if validated in this study.

In terms of potential risks or burdens involved, there will be no physical risks incurred by participation in the study. Recruited women will not be expected to have any additional visits to the hospital during the study, over and above usual care. The investigators are aware that when conducting a study of anxiety symptoms, it could potentially identify a woman with an undiagnosed mental health condition, issues of self-harm or potential harm to others. The principal investigator will check the survey responses regularly and will highlight any responses which are of serious concern. The investigator will then contact the woman directly to discuss her responses. The participant will be encouraged to see the General Practitioner (GP) if deemed necessary. If the participant does not wish to see the GP or there is persistent concern from the local researcher the confidentiality clause may need to be broken in the interest of safety of the participant and others. The local researcher will then contact the GP directly after informing the participant of their intended actions, to report these concerns.It is possible that the participants will not perceive any individual benefit from participating in this study. It is possible that the women will not perceive any individual benefit from participating in this study.

A statistician will be consulted to assist in analysis of the data collected from the study.

To calculate the sample sizes, power calculations were performed on the HADS scale. Puhan et al (2008) report the minimal important difference in HADS scores is 1.5 units for a significance level of 0.05 and a statistical power of 80% when considering an intervention. Based upon this assumption and a common standard deviation of 4 points, 125 women are needed for each group (total 250 women). A drop-out rate of 10% is anticipated.

The following statistical analyses will be performed:

Descriptive statistics will be used to compare the two groups in terms of baseline demographic characteristics. Continuous variables normally distributed will be described reporting mean and standard deviation, otherwise median and interquartile range will be used. Categorical variables will be reported with frequency tables. To compare HADS scores between groups I and II, the t-test will be performed for continuous variables normally distributed, otherwise the Mann-Whitney U test will be used. The Chi-squared test will be used for categorical variables.

A statistically significant difference will be considered as a p-value <0.05. The data will be checked for abnormalities, spurious and missing data. These will be coded separately and treated accordingly. Analyses will be carried out using Stata statistical software, Release 14 (StataCorp, College Station, TX).

Throughout the study (and afterwards), the research investigators will welcome inspections and monitoring of the conduct of the research to ensure that the quality of the research is upheld and that the agreed practice is being adhered to. This includes offering direct access to any documents.

Data will be stored on secure computers at the specific hospital conducting the study using password protected access to databases. Hard copy data (consent and registration forms) will be stored within the unit site files which will be kept in secure areas.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years+
* Diagnosis of IPUVI on initial ultrasound

Exclusion Criteria:

* Current mental health condition (anxiety, depression, eating disorder). The condition will be considered current if it has required one or more consultations with a medical professional (including a psychologist) over the past 6 months (women with past mental health condition will not be excluded)
* The patient is planning a termination
* Multiple order pregnancies
* Women who in the opinion of the researcher by virtue of language or learning impairment would be unable to give fully informed consent to the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
A change in self-reported psychological well-being from diagnosis to follow-up between the two groups. | 14 days
  To assess and compare if there is any significant difference in symptoms of anxiety and depression during the uncertain period, as measured by the Hospital and Anxiety Depression Score in the two groups of women all diagnosed with IPUVI. The two groups will be; 1) women randomised to receive the prediction tool and 2) women randomised to not receive the prediction tool.
  2. To assess and compare whether the symptoms of anxiety and depression in the two groups of women change over three defined time points: immediately after the initial ultrasound/ diagnosis, at 72 hours post ultrasound and immediately prior to the follow-up ultrasound at 14 days.
  The questionnaire has two components, one relating to anxiety symptoms (HADS-A) and one relating to depressive symptoms (HADS-D). Each component comprises seven statements. Each statement is scored 0-3 yielding a total of 0-21 points for each component.

SECONDARY OUTCOMES:
Patient Experience of the prediction tool | 14 days
  3. To assess the patient experience during the study period by applying a self-reported experience questionnaire on the acceptability and perceived usefulness of the prediction tool, in those women who receive it. The questionnaire has been developed by the study investigators using modified versions of the Technology Acceptance Model by Davis et al, 1989.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Bottomley, MRCOG MD, Study Chair — Chelsea and Westminster NHS Foundation Trust; Kim K Lawson, MBChB, Principal Investigator — Chelsea and Westminster NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bottomley C, Van Belle V, Mukri F, Kirk E, Van Huffel S, Timmerman D, Bourne T. The optimal timing of an ultrasound scan to assess the location and viability of an early pregnancy. Hum Reprod. 2009 Aug;24(8):1811-7. doi: 10.1093/humrep/dep084. Epub 2009 Apr 10. PMID 19363041
- [Background] Davison AZ, Appiah A, Sana Y, Johns J, Ross JA. The psychological effects and patient acceptability of a test to predict viability in early pregnancy: a prospective randomised study. Eur J Obstet Gynecol Reprod Biol. 2014 Jul;178:95-9. doi: 10.1016/j.ejogrb.2014.04.002. Epub 2014 Apr 18. PMID 24837026
- [Background] Richardson A, Raine-Fenning N, Deb S, Campbell B, Vedhara K. Anxiety associated with diagnostic uncertainty in early pregnancy. Ultrasound Obstet Gynecol. 2017 Aug;50(2):247-254. doi: 10.1002/uog.17214. Epub 2017 Jun 27. PMID 27484256
- [Background] Bottomley C, Van Belle V, Kirk E, Van Huffel S, Timmerman D, Bourne T. Accurate prediction of pregnancy viability by means of a simple scoring system. Hum Reprod. 2013 Jan;28(1):68-76. doi: 10.1093/humrep/des352. Epub 2012 Oct 30. PMID 23111205
- [Background] Bottomley C, Van Belle V, Pexsters A, Papageorghiou AT, Mukri F, Kirk E, Van Huffel S, Timmerman D, Bourne T. A model and scoring system to predict outcome of intrauterine pregnancies of uncertain viability. Ultrasound Obstet Gynecol. 2011 May;37(5):588-95. doi: 10.1002/uog.9007. PMID 21520315
- [Background] Lok IH, Neugebauer R. Psychological morbidity following miscarriage. Best Pract Res Clin Obstet Gynaecol. 2007 Apr;21(2):229-47. doi: 10.1016/j.bpobgyn.2006.11.007. Epub 2007 Feb 20. PMID 17317322
- [Background] Farren J, Jalmbrant M, Ameye L, Joash K, Mitchell-Jones N, Tapp S, Timmerman D, Bourne T. Post-traumatic stress, anxiety and depression following miscarriage or ectopic pregnancy: a prospective cohort study. BMJ Open. 2016 Nov 2;6(11):e011864. doi: 10.1136/bmjopen-2016-011864. PMID 27807081
- [Background] Guha S, Van Belle V, Bottomley C, Preisler J, Vathanan V, Sayasneh A, Stalder C, Timmerman D, Bourne T. External validation of models and simple scoring systems to predict miscarriage in intrauterine pregnancies of uncertain viability. Hum Reprod. 2013 Nov;28(11):2905-11. doi: 10.1093/humrep/det342. Epub 2013 Aug 26. PMID 23980057

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT03264170/Prot_SAP_000.pdf